CLINICAL TRIAL: NCT06365060
Title: Screening for AL Amyloidosis in Smoldering Multiple Myeloma
Status: Recruiting | Type: Observational
Sponsor: Tufts Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 00003143; R01CA279808 (NIH)
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Smoldering Multiple Myeloma
Keywords: SMM; AL Amyloidosis
MeSH Terms: conditions — Smoldering Multiple Myeloma; Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cDNA derived from bone marrow CD138-selected plasma cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In this multicenter study, we will recruit 400 patients 40 years of age or older at 15 centers with a diagnosis of smoldering multiple myeloma (SMM), a group of patients for whom standard of care is observation not treatment. The main goal of this study is to screen for the diagnosis of light-chain amyloidosis (AL) before the onset of symptomatic disease and to develop a training set for a likelihood algorithm.

DETAILED DESCRIPTION:
This study is based on results from two prior studies in which 4 of 36 patients with SMM and none of 14 patients with MGUS were found to have AL. The hypothesis that we test with this protocol is that patients with (1) a pre-existing diagnosis of SMM, (2) free light chain (FLC) abnormalities, (3) IGLV genes associated with AL,(4) t(11;14) or gain 1q, and (5) NT-proBNP > 332pg/mL will have undiagnosed AL or risk of progression to AL. We will study the potential for SMM, the FLC screen, AL-related IGLV gene use, t(11;14) or gain 1q cytogenetic abnormalities, and NT-proBNP > 332pg/mL to be the variables in a likelihood algorithm for AL.

ELIGIBILITY:
Inclusion Criteria:

* Patients 40 years of age and older
* diagnosed with either Smoldering Multiple Myeloma or a Monoclonal Gammopathy
* dFLC greater than 23 mg/L
* abnormal FLC ratio
* If the patient has an eGFR less than 50 mL/min/1.73m2, the FLC ratio is inconsequential. The patient only needs to meet the age and dFLC criterion.

Exclusion Criteria:

* Patients younger than 40 years of age are not eligible
* Patients with a previous finding of amyloid in other biopsies will not be included
* Adults unable to consent are not eligible, including the cognitively impaired Pregnant women, pregnant minors, minors (i.e., individuals who are not yet adults), wards of the state, non-viable neonates, neonates of uncertain viability, and prisoners are not eligible

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Smoldering Multiple Myeloma patients.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2029-02-27 (Estimated); Study Completion 2029-02-27 (Estimated)

PRIMARY OUTCOMES:
Creating a network to enroll patients on a collaborative study requiring marrow and blood specimens, to collect data for a training set of likelihood statistics and to plan a future validation study. | 5 years
  With a 15-center network covering 12 states and almost 45% of the US population, we will evaluate 400 SMM patients > 40 years old who pass FLC criteria using standard of care tests including NT-proBNP and clinical marrow specimens evaluated for the presence of t(11;14) and gain1q. Marrow cells will be processed by NGS for clonal IGLV gene identification. With the training data obtained, we will use existing statistical modeling techniques to generate a statistical algorithm for identifying undiagnosed cases of AL and assessment of risk of AL, and to plan a validation study testing the training model. We will also investigate a role for the novel biomarker clusterin (Clu) as an indicator of risk of AL in SMM patients; preliminary work indicates that Clu is significantly lower in AL than in SMM patients.
Validating an NGS assay that identifies IGLV genes in clonal plasma cells | 5 years
  All subjects will have their clonal IGLV genes identified by NGS enabling the creation and validation of a laboratory developed test in a precision medicine laboratory that is certified under regulations of the Clinical Laboratory Improvement Amendments of 1988 (CLIA). Approval for this laboratory developed test for both κ and λ IGVL genes will permit providers, patients and researchers to use the test in decision-making to care for monoclonal gammopathy patients. We will also investigate the exploratory objective of defining the alterations in sequence in AL and non-AL FLC derived from the same IGLV germline gene.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - University of Alabama Hospital, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Cleveland Clinic Florida, Weston Hospital, Weston, Florida
  - Tufts Medical Center, Boston, Massachusetts
  - Columbia University Irving Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Atrium Health Levine Cancer Institute, Charlotte, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Durham, North Carolina
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - UT Southwestern, Harold C. Simmons Comprehensive Cancer Center, Dallas, Texas
  - University of Utah, Huntsman Cancer Hospital, Salt Lake City, Utah
  - VCU Medical Center, Richmond, Virginia

REFERENCES:
- [Background] Avalos M, Pouyes H, Grandvalet Y, Orriols L, Lagarde E. Sparse conditional logistic regression for analyzing large-scale matched data from epidemiological studies: a simple algorithm. BMC Bioinformatics. 2015;16 Suppl 6(Suppl 6):S1. doi: 10.1186/1471-2105-16-S6-S1. Epub 2015 Apr 17. PMID 25916593
- [Background] Bodi K, Prokaeva T, Spencer B, Eberhard M, Connors LH, Seldin DC. AL-Base: a visual platform analysis tool for the study of amyloidogenic immunoglobulin light chain sequences. Amyloid. 2009 Mar;16(1):1-8. doi: 10.1080/13506120802676781. PMID 19291508
- [Background] Bujang MA, Adnan TH. Requirements for Minimum Sample Size for Sensitivity and Specificity Analysis. J Clin Diagn Res. 2016 Oct;10(10):YE01-YE06. doi: 10.7860/JCDR/2016/18129.8744. Epub 2016 Oct 1. PMID 27891446
- [Background] Comenzo RL, Wally J, Kica G, Murray J, Ericsson T, Skinner M, Zhang Y. Clonal immunoglobulin light chain variable region germline gene use in AL amyloidosis: association with dominant amyloid-related organ involvement and survival after stem cell transplantation. Br J Haematol. 1999 Sep;106(3):744-51. doi: 10.1046/j.1365-2141.1999.01591.x. PMID 10468868
- [Background] Comenzo RL, Zhang Y, Martinez C, Osman K, Herrera GA. The tropism of organ involvement in primary systemic amyloidosis: contributions of Ig V(L) germ line gene use and clonal plasma cell burden. Blood. 2001 Aug 1;98(3):714-20. doi: 10.1182/blood.v98.3.714. PMID 11468171
- [Background] Chaulagain CP, Comenzo RL. How we treat systemic light-chain amyloidosis. Clin Adv Hematol Oncol. 2015 May;13(5):315-24. PMID 26352777
- [Background] Dasari S, Theis JD, Vrana JA, Meureta OM, Quint PS, Muppa P, Zenka RM, Tschumper RC, Jelinek DF, Davila JI, Sarangi V, Kurtin PJ, Dogan A. Proteomic detection of immunoglobulin light chain variable region peptides from amyloidosis patient biopsies. J Proteome Res. 2015 Apr 3;14(4):1957-67. doi: 10.1021/acs.jproteome.5b00015. Epub 2015 Mar 20. PMID 25734799
- [Background] Dispenzieri A, Kyle RA, Katzmann JA, Therneau TM, Larson D, Benson J, Clark RJ, Melton LJ 3rd, Gertz MA, Kumar SK, Fonseca R, Jelinek DF, Rajkumar SV. Immunoglobulin free light chain ratio is an independent risk factor for progression of smoldering (asymptomatic) multiple myeloma. Blood. 2008 Jan 15;111(2):785-9. doi: 10.1182/blood-2007-08-108357. Epub 2007 Oct 17. PMID 17942755
- [Background] Dubrey SW, Cha K, Anderson J, Chamarthi B, Reisinger J, Skinner M, Falk RH. The clinical features of immunoglobulin light-chain (AL) amyloidosis with heart involvement. QJM. 1998 Feb;91(2):141-57. doi: 10.1093/qjmed/91.2.141. PMID 9578896
- [Background] Kourelis TV, Kumar SK, Go RS, Kapoor P, Kyle RA, Buadi FK, Gertz MA, Lacy MQ, Hayman SR, Leung N, Dingli D, Lust JA, Lin Y, Zeldenrust SR, Rajkumar SV, Dispenzieri A. Immunoglobulin light chain amyloidosis is diagnosed late in patients with preexisting plasma cell dyscrasias. Am J Hematol. 2014 Nov;89(11):1051-4. doi: 10.1002/ajh.23827. Epub 2014 Sep 2. PMID 25111004
- [Background] Kyle RA, Rajkumar SV. Monoclonal gammopathy of undetermined significance and smoldering multiple myeloma. Curr Hematol Malig Rep. 2010 Apr;5(2):62-9. doi: 10.1007/s11899-010-0047-9. PMID 20425398
- [Background] Kyle RA, Remstein ED, Therneau TM, Dispenzieri A, Kurtin PJ, Hodnefield JM, Larson DR, Plevak MF, Jelinek DF, Fonseca R, Melton LJ 3rd, Rajkumar SV. Clinical course and prognosis of smoldering (asymptomatic) multiple myeloma. N Engl J Med. 2007 Jun 21;356(25):2582-90. doi: 10.1056/NEJMoa070389. PMID 17582068
- [Background] Larsen JT, Kumar SK, Dispenzieri A, Kyle RA, Katzmann JA, Rajkumar SV. Serum free light chain ratio as a biomarker for high-risk smoldering multiple myeloma. Leukemia. 2013 Apr;27(4):941-6. doi: 10.1038/leu.2012.296. Epub 2012 Oct 16. PMID 23183428
- [Background] Perfetti V, Casarini S, Palladini G, Vignarelli MC, Klersy C, Diegoli M, Ascari E, Merlini G. Analysis of V(lambda)-J(lambda) expression in plasma cells from primary (AL) amyloidosis and normal bone marrow identifies 3r (lambdaIII) as a new amyloid-associated germline gene segment. Blood. 2002 Aug 1;100(3):948-53. doi: 10.1182/blood-2002-01-0114. PMID 12130507
- [Background] Perfetti V, Palladini G, Casarini S, Navazza V, Rognoni P, Obici L, Invernizzi R, Perlini S, Klersy C, Merlini G. The repertoire of lambda light chains causing predominant amyloid heart involvement and identification of a preferentially involved germline gene, IGLV1-44. Blood. 2012 Jan 5;119(1):144-50. doi: 10.1182/blood-2011-05-355784. Epub 2011 Nov 8. PMID 22067386
- [Background] Rajkumar SV, Kyle RA, Therneau TM, Melton LJ 3rd, Bradwell AR, Clark RJ, Larson DR, Plevak MF, Dispenzieri A, Katzmann JA. Serum free light chain ratio is an independent risk factor for progression in monoclonal gammopathy of undetermined significance. Blood. 2005 Aug 1;106(3):812-7. doi: 10.1182/blood-2005-03-1038. Epub 2005 Apr 26. PMID 15855274
- [Background] Tahir UA, Doros G, Kim JS, Connors LH, Seldin DC, Sam F. Predictors of Mortality in Light Chain Cardiac Amyloidosis with Heart Failure. Sci Rep. 2019 Jun 12;9(1):8552. doi: 10.1038/s41598-019-44912-x. PMID 31189919
- [Background] Zhou P, Comenzo RL, Olshen AB, Bonvini E, Koenig S, Maslak PG, Fleisher M, Hoffman J, Jhanwar S, Young JW, Nimer SD, Boruchov AM. CD32B is highly expressed on clonal plasma cells from patients with systemic light-chain amyloidosis and provides a target for monoclonal antibody-based therapy. Blood. 2008 Apr 1;111(7):3403-6. doi: 10.1182/blood-2007-11-125526. Epub 2008 Jan 23. PMID 18216299
- [Background] Zhou P, Hoffman J, Landau H, Hassoun H, Iyer L, Comenzo RL. Clonal plasma cell pathophysiology and clinical features of disease are linked to clonal plasma cell expression of cyclin D1 in systemic light-chain amyloidosis. Clin Lymphoma Myeloma Leuk. 2012 Feb;12(1):49-58. doi: 10.1016/j.clml.2011.09.217. Epub 2011 Nov 18. PMID 22100494
- [Background] Zhou P, Ma X, Iyer L, Chaulagain C, Comenzo RL. One siRNA pool targeting the lambda constant region stops lambda light-chain production and causes terminal endoplasmic reticulum stress. Blood. 2014 May 29;123(22):3440-51. doi: 10.1182/blood-2013-10-535187. Epub 2014 Apr 10. PMID 24723680
- [Background] Hutchison CA, Harding S, Hewins P, Mead GP, Townsend J, Bradwell AR, Cockwell P. Quantitative assessment of serum and urinary polyclonal free light chains in patients with chronic kidney disease. Clin J Am Soc Nephrol. 2008 Nov;3(6):1684-90. doi: 10.2215/CJN.02290508. PMID 18945993
- [Background] Singh G. Serum Free Light Chain Assay and kappa/lambda Ratio Performance in Patients Without Monoclonal Gammopathies: High False-Positive Rate. Am J Clin Pathol. 2016 Aug;146(2):207-14. doi: 10.1093/ajcp/aqw099. PMID 27473738